CLINICAL TRIAL: NCT04748887
Title: Chronic Obstructive Pulmonary Disease in Non Smokers:Role of Oxidative Stress
Brief Title: Oxidative Stress Markers in COPD
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, zainab hassan saeed, principle investigator ,faculty of medicine,department of chest diseases,Minia University, Minia University
Other Study IDs: oxidative stress
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Role of Oxidative Stress in COPD
Keywords: COPD , oxidative stress, Superoxide Dismutase
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Superoxide Dismutase; Malondialdehyde

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nonsmokers copd cases ,: Fourty subjects of COPD who are non-smokers or stopped smoking for more than 6 months
  Interventions: Other: oxidative stess markers
- non smokers healthy control: Thirty subjects of non smokers healthy control
  Interventions: Other: oxidative stess markers

INTERVENTIONS:
Other: oxidative stess markers — markers of oxidative stress , Superoxide Dismutase (SOD) and Malondialdehyde (MDA) by ( ELISA Kit SinoGeneClon Biotech Co.,Ltd Catalog No : SG- 10188) .
  Other Names: Superoxide Dismutase (SOD) and Malondialdehyde (MDA)

SUMMARY:
Background:Striking feature of Chronic obstructive pulmonary disease (COPD) is its inability to resolve after cigarette smoke exposure has ended, which has contributed to the possibility that the disease could also be driven by other endogenous causes, such as autoimmunity or chronic infection . Many of the pathogenetic pathways involved in COPD and its development tend to be driven by oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* 1-Forty subjects of COPD who are non-smokers or stopped smoking for more than 6 months Based on the Global Initiative for Chronic Obstructive Lung Disease guidelines, COPD was diagnosed.9 2- Thirty subjects of non smokers healthy control

Exclusion Criteria:

* Patients of:

  1. Acute exacerbation, at the time of the study, of COPD.
  2. Any obvious abnormal lung parenchymal lesions.
  3. Lung cancer.
  4. Congestive heart failure.
  5. current smokers
  6. Drugs e.g anti-inflammatory , steroids ,analgesics, insulin , antineoplastic, antipsychotic drugs in the previous 2 weeks before the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Forty subjects of COPD who are non-smokers or stopped smoking for more than 6 months Based on the Global Initiative for Chronic Obstructive Lung Disease guidelines, COPD was diagnosed.9 2- Thirty subjects of non smokers healthy control
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
oxidative stress markers in non smokers COPD compared to healthy control | 1month
  markers of oxidative stress , Superoxide Dismutase (SOD) and Malondialdehyde (MDA) by ( ELISA Kit SinoGeneClon Biotech Co.,Ltd Catalog No : SG- 10188) .

CONTACTS AND LOCATIONS:
Overall Officials: zainab H Saeed, MD, Principal Investigator — MD chest diseases
Locations (1):
- Minia University Hospital, Multiple Locations, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No